CLINICAL TRIAL: NCT06054633
Title: Efficacy and Safety of Oral L-Arginine for Pain Relief in Knee Osteoarthritis: a Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: L-arginine for Knee Osteoarthritis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Massachusetts General Hospital (Other); School of Medicine, University of Nottingham (Unknown); Memorial University of Newfoundland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20230608
Record Dates: First submitted 2023-09-17; First posted 2023-09-26 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; L-arginine; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral L-arginine (Active Comparator): Participants in the intervention arm will receive oral L- arginine tablets, 2 g three times daily
  Interventions: Dietary Supplement: L-arginine tablet
- Placebo (Placebo Comparator): The control group will receive an identical inert placebo tablet, three times daily
  Interventions: Dietary Supplement: Placebo tablet

INTERVENTIONS:
Dietary Supplement: L-arginine tablet — L-arginine, 2 g, three times daily, for 12 weeks
  Arms: Oral L-arginine
Dietary Supplement: Placebo tablet — Identical inert placebo, three times daily, for 12 weeks
  Arms: Placebo

SUMMARY:
This study will examine the pain-relief efficacy and safety of L-arginine in knee OA patients.

DETAILED DESCRIPTION:
Pain is the dominant symptom of knee osteoarthritis (KOA). The main management goal for people with KOA is to control pain without increasing treatment-related adverse effects (AEs). However, the commonly prescribed systemic analgesics have safety concerns, such as increased risk of cardiovascular and gastrointestinal AEs. Therefore, it is urgent to develop safe and effective treatment options.

L-arginine is one of the most commonly used oral nutritional supplements that has been widely used in patients with peripheral arterial disease, cystic fibrosis, and pregnant women with high risk of pre-eclampsia. The supplement has a high safety profile. Previous case-control and cross-sectional studies have found plasma L-arginine levels were lower in patients with knee OA than controls, suggesting that arginine deficiency may increase the risk of OA. The investigators previously observed an inverse dose-response relationship between levels of serum L-arginine and the risk of incident symptomatic KOA. Additionally, the investigators demonstrated that intra-articular injection of L-arginine solution relieved pain symptoms in a surgical rat model of OA. However, there is a paucity of high-quality clinical evidence on the effect of intake of L-arginine supplement on pain relief among patients with symptomatic KOA.

The investigators propose to conduct a randomized, double-blind, placebo-controlled trial to examine the efficacy and safety of oral L-arginine in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 80 years.
2. Knee OA according to the American College of Rheumatology (ACR) clinical criteria.
3. Knee pain lasting 3 months or longer and a score of 7 or greater on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale (standardized to range from 0-20).
4. Kellgren-Lawrence (KL) grade 2 or 3.
5. Willing to and able to provide written informed consent.

Exclusion Criteria:

1. Any use of NSAIDs or other analgesics in the past two weeks.
2. History of injections of corticosteroids in the past three months or hyaluronic acid in the past 6 months in the index knee.
3. History of arthroscopy or open surgery in the index knee in the past 12 months.
4. History of a knee replacement in the index knee or planning to receive such a procedure within 3 months.
5. History of a severe injury in the index knee.
6. Pain in the index knee caused by inflammatory, autoimmune, neoplastic diseases or other diseases.
7. Abnormal liver or kidney functions, as defined by alanine transaminase or aspartate aminotransferase >two times the upper limit of normal, or blood urea nitrogen or serum creatinine >two times the upper limit of normal.
8. Severe respiratory diseases.
9. History of coronary artery disease and heart failure.
10. Uncontrolled hypertension or diabetes mellitus.
11. Diagnosis of malignant tumors.
12. Pregnant or contemplating pregnancy or breast-feeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score. | Baseline, Week 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of WOMAC have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.

SECONDARY OUTCOMES:
Change From Baseline in WOMAC pain score. | Baseline, Weeks 2, 4 and 8
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of WOMAC have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Change From Baseline in Knee pain on a visual analogue scale (VAS). | Baseline, Weeks 2, 4, 8 and 12
  Knee pain will be graded by a VAS from 0 to 100 mm, with 0 indicating "No pain" and 100 indicating "Worst possible pain".
Change From Baseline in WOMAC total score. | Baseline, Weeks 2, 4, 8 and 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of this index have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Change From Baseline in Change From Baseline in WOMAC stiffness score. | Baseline, Weeks 2, 4, 8 and 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of WOMAC have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Change From Baseline in WOMAC function score. | Baseline, Weeks 2, 4, 8 and 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of WOMAC have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Change From Baseline in Patient global assessment of osteoarthritis (PGA-OA) score. | Baseline, Weeks 2, 4, 8 and 12
  PGA-OA score will be assessed using a 100 mm visual analogue scale (higher is worse).
Change From Baseline in SF-12 questionnaire score. | Baseline, Weeks 2, 4, 8 and 12
  The SF-12 Quality of Life questionnaire includes 8 multi-item domains (physical function, social function, role-emotional, role-physical, bodily pain, general health, mental health, and vitality). These can be combined into 2 summary measures (physical and mental component summary measures).
Change From Baseline in Timed Up and Go Test (TUG). | Baseline, Weeks 4, 8 and 12
  TUG is a functional performance measure specifically studied in persons with OA of the hip and knee, which directly evaluates an individual's ability to transfer, ambulate, and maintain balance during transitions. The TUG assesses the time it takes participants to get up from a standard-height chair, walk 3 m, turn and return to the chair, and sit down again. The TUG has good interrater and intrarater reliability and validity for functional testing in older adults.
Change From Baseline in Chair-stand Test. | Baseline, Weeks 4, 8 and 12
  The chair-stand test will use a standard chair with a 47-cm seat height. Participants start the test seated, with arms crossed over the chest, and are instructed to rise to a full stand and return to the initial seated position as many times as possible in 30 seconds. The total number of completed chair stands is averaged across two trials and used for analysis. A greater number of chair stand repetitions is interpreted as better performance.
Change From Baseline in Ultrasound-assessed knee synovitis. | Baseline, Week 12
  Both knees will be assessed with the participant supine and the knee in 30° flexion. The suprapatellar bursa will be scanned according to the Outcome Measures in Rheumatology (OMERACT) atlas. Maximal depth of effusion and synovial thickness will be measured in millimeters. Power Doppler signal observed in the synovial membrane in both longitudinal and transverse planes will be scored using a semi-quantitative grading system, from 0 to 3 (0 = absent, 1 = mild, 2 = moderate, 3 = marked or severe).
Rescue medicine consumption. | Weeks 2, 4, 8 and 12
  The consumption of rescue medication will be recorded at each visit and in the daily logs.
Change From Baseline in Level of C-reactive protein (CRP). | Baseline, Weeks 4, 8 and 12
  The blood samples will be collected in the morning after an overnight fast at baseline and the following visits to measure the level of CRP in serum.
Change From Baseline in Microbiota diversity and composition. | Baseline, Weeks 4, 8 and 12
  Stool and saliva samples will be collected at baseline and the following visits. Microbial diversity will be quantified via the Shannon diversity index (α diversity) and unweighted Unifrac distance (β diversity), and microbiota composition will be identified on different levels, including phylum, family, and genus.
Incidence of adverse events and serious adverse events. | Weeks 2, 4, 8 and 12
  Adverse events and serious adverse events will be measured and recorded.

OTHER OUTCOMES:
Change From Baseline in Short Physical Performance Battery (SPPB) scores. | Baseline, Weeks 4, 8 and 12
  The SPPB is a standardized, reproducible measure of global physical function validated in frail older persons that predicts a wide range of clinical outcomes. It has 3 components: a standing balance test, gait speed (4-meter walk) test, and strength test (time to complete 5 chair rises). Each component is scored 0-4 for a total score ranging from 0-12, where lower scores indicate more severe physical dysfunction.
Change From Baseline in Grip strength. | Baseline, Weeks 4, 8 and 12
  The grip strength of the participants' dominant hand will be measured using a calibrated Jamar dynamometer with the participants in the sitting position (Patterson Medical, Ltd., Nottinghamshire, UK). Three grip strength measurements will be taken at 10 s intervals, and the maximum value of the three measurements will be used as the participant's final grip strength.
Change From Baseline in Bone mineral density (BMD). | Baseline, Week 12
  A trained technician will measure the BMD of all participants. The total body BMD and multiple site-specific BMD (i.e., the lumbar spine, pelvis, trunk, femoral neck, trochanteric, and ward's triangle) will be all measured. The dual-energy X-ray absorptiometry (DXA) scan results are reported as absolute values of BMD (g/cm2). The same DXA machine will be used for all participants. All technicians will receive training to ensure the reproducibility of the BMD measures.
Change From Baseline in DXA-based whole-body muscle mass. | Baseline, Week 12
  Body composition assessment provides insights into the nutritional status and functional capacity. It helps understand nutrition in the developmental origins of health and disease and in monitoring therapeutic interventions. The whole body muscle mass will be measured using DXA.
Change From Baseline in DXA-based whole body fat mass. | Baseline, Week 12
  Body composition assessment provides insights into the nutritional status and functional capacity. It helps understand nutrition in the developmental origins of health and disease and in monitoring therapeutic interventions. The whole body fat mass will be measured using DXA.
Change From Baseline in pressure pain threshold (PPT). | Baseline, Weeks 4, 8 and 12
  PPT measures sensitivity to pain evoked by mechanical stimulation of nociceptors. PPT will be assessed at the center of patellar in the index knee and at the distal radioulnar joint (right side unless contraindicated) by applying an algometer (1 cm2 rubber tip; Wagner, FDIX25) at a rate of 0.5 kg/s, with the calculation of averaging three trials at each site.
Change From Baseline in mechanical temporal summation (mTS). | Baseline, Weeks 4, 8 and 12
  Mechanical temporal summation (mTS) measures an augmented response to repetitive mechanical stimulation. mTS will be assessed using a weighted 60 g von Frey monofilament at the center of patellar in the index knee and at the distal radioulnar joint (right side unless contraindicated). Subjects first provided a numerical pain rating to a trial of four stimulations. Subsequently, the monofilament was applied repeatedly over the skin of the same site at a frequency of 1 Hz for 30 s. Subjects provided a pain rating at the completion of the train of 30 simulations, and 15 s post stimulation. Temporal summation was defined as being present when, compared with the initial trial, the subject reported increased pain following the repeated mechanical stimulation at the site being tested. If there is no difference between the two trials, then the participant is not defined as temporal summation.
Change From Baseline in Hospital Anxiety and Depression Scale (HADS). | Baseline, Weeks 4, 8 and 12
  HADS is a self-report scale and consists of 14 items, 7 of which investigate depression and 7 anxiety symptoms, providing a score of 0 to 21 for each domain, where higher scores equal greater involvement of either anxiety or depression. The purpose of the scale is not to make a diagnosis. It is to determine the risk group by screening for anxiety and depression in a short time in patients with physical illness. In addition, the scale can be used to evaluate the change in the emotional status of patients.
Change From Baseline in PainDETECT Questionnaire (PD-Q). | Baseline, Weeks 4, 8 and 12
  The PD-Q includes three questions about knee pain intensity rated via NRSs ("no pain" (score 0) to "worst pain possible" (score 10)), pain course pattern rated via a diagram displaying four possible pain course patterns (scored -1 to 2 depending on which pain course pattern is selected), a question about pain radiation (answered yes/no, and scored 2 or 0 respectively), and seven questions about somatosensory phenomena each rated on 6-point Likert scales ("never" (score 0) to "very strongly" (score 5)). Total scores are obtained by summing scores for all items, ranging from 0 to 38. Higher scores indicate more neuropathic-like symptoms. Scores of ≤12 indicate pain is unlikely to be neuropathic and scores of ≥19 suggest pain is likely to have a neuropathic component. Scores ≥13 and ≤18 indicate uncertain results and the possibility of a neuropathic component.

CONTACTS AND LOCATIONS:
Overall Officials: Guanghua Lei, MD, PhD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No